CLINICAL TRIAL: NCT01856114
Title: A Preliminary Study of Prophylactic Fentanyl Buccal Tablets (FBT) for Exercise Induced Breakthrough Dyspnea
Brief Title: Fentanyl Buccal Tablets for Exercise Induced Breakthrough Dyspnea
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: Teva Pharmaceuticals USA (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2013-0043; NCI-2014-01033 (Registry Identifier: NCI CTRP)
Record Dates: First submitted 2013-05-14; First posted 2013-05-17 (Estimated); Results first posted 2020-09-16 (Actual); Last update posted 2020-09-16 (Actual); Status verified 2020-09

CONDITIONS: Advanced Cancers
Keywords: Advanced Cancers; Cancer with evidence of active disease; Exercise induced breakthrough dyspnea; Shortness of breath; Fentanyl Buccal Tablets; FBT; Placebo; Walk tests; Questionnaires; Surveys
MeSH Terms: conditions — Dyspnea | interventions — Surveys and Questionnaires

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Fentanyl Buccal Tablet (Experimental): After a six minute walk test, participant will sit down and rest for up to 1 hour. They will then be given a Fentanyl tablet to put in between upper gum and cheek. Study physician will determine the morphine equivalent daily dose (MEDD) in real time using standardized equianalgesic ratios. Based on clinical practice and similarly to the dose used for breakthrough pain, an FBT dose equivalent to 20-50% of the MEDD used. After 30 minutes, participant asked about any side effects they may be having, and repeat the walking test. During each walk test, participant asked 6 times how hard it is to catch their breath. The total distance walked will also be recorded. Completion of two questionnaires at beginning of study visit. It should take about 10 minutes to complete. At the end of study visit, completion of last questionnaire. It should take about 5 minutes to complete the questionnaire.
  Interventions: Drug: Fentanyl Buccal Tablet; Behavioral: Questionnaires
- Placebo Buccal Tablet (Placebo Comparator): After a six minute walk test, participant will sit down and rest for up to 1 hour. They will then be given a Placebo tablet to put in between upper gum and cheek. After 30 minutes, participant asked about any side effects they may be having, and repeat the walking test. During each walk test, participant asked 6 times how hard it is to catch their breath. The total distance walked will also be recorded. Completion of two questionnaires at beginning of study visit. It should take about 10 minutes to complete. At the end of study visit, completion of last questionnaire. It should take about 5 minutes to complete the questionnaire.
  Interventions: Other: Placebo Buccal Tablet; Behavioral: Questionnaires

INTERVENTIONS:
Drug: Fentanyl Buccal Tablet — Fentanyl buccal tablet given to put in between upper gum and cheek one hour after a six minute walk test.
  Arms: Fentanyl Buccal Tablet
Other: Placebo Buccal Tablet — Placebo buccal tablet given to put in between upper gum and cheek one hour after a six minute walk test.
  Arms: Placebo Buccal Tablet
Behavioral: Questionnaires — Completion of two questionnaires at beginning of study visit. It should take about 10 minutes to complete. At the end of study visit, completion of last questionnaire. It should take about 5 minutes to complete the questionnaire.
  Other Names: Surveys

SUMMARY:
The goal of this clinical research study is to learn if fentanyl can change perception of shortness of breath in cancer patients. Researchers also want to learn if the study drug can help to improve your physical function. In this study, fentanyl will be compared to a placebo.

Fentanyl is commonly used for treatment of cancer pain.

A placebo is not a drug. It looks like the study drug but is not designed to treat any disease or illness. It is designed to be compared with a study drug to learn if the study drug has any real effect.

DETAILED DESCRIPTION:
Study Groups:

If you are found to be eligible to take part in this study, you will be randomly assigned (as in the flip of a coin) to either receive fentanyl or placebo. You will have an equal chance of being assigned to either group. Neither you nor the study staff will know if you are receiving the study drug or the placebo. However, if needed for your safety, the study staff will be able to find out what you are receiving.

Study Visit:

During your study visit, the study staff will collect information from your medical record about your age, sex, race, disease type, how well you are able to perform the normal activities of daily living, any drugs you are taking, and possible causes of shortness of breath.

You will complete 2 questionnaires. One (1) of them will have questions about any breathing symptoms you may be having, and the other asks about any other symptoms you may be having. It should take about 10 minutes to complete these questionnaires.

The study staff will then record your vital signs (heart rate, breathing rate, and the level of air breathed out using a measuring device that will be clipped onto your finger). You will also be asked how hard it is to catch your breath and to rate your level of tiredness.

You will then walk back and forth in an indoor corridor for up to 6 minutes. This is called a walk test. You may slow down, stop, and rest at any time you need to.

After that, you will sit down and rest for up to 1 hour. During this time, the study drug/placebo will be prepared and you may be asked several times how hard it is to catch your breath.

You will then be given a study drug/placebo tablet to put it in between your upper gum and cheek. You will then wait for another 30 minutes, be asked about any side effects you may be having, and repeat the walking test. Then the study staff will ask you again about any side effects you may be having, your level of tiredness, and how hard it is to catch your breath. Your vital signs will also be measured.

During each walk test, you will be asked 6 times how hard it is to catch your breath. How often you stopped and for how long will be recorded. The total distance you walked will also be recorded.

After each walk test, you will also be asked to complete 4 tests of your mental abilities, including finger tapping, simple mathematics questions (addition, subtraction, multiplication, division), recall of numbers, and recall of objects. It should take 15 minutes to complete these tests.

At the end of the study visit, you will fill out 1 questionnaire that asks if you think the study drug/placebo is helping you, how satisfied you are with the study, and which treatment you think you received. It should take about 5 minutes to complete the questionnaire.

Length of Study:

Your active participation in this study is over after you complete the last questionnaire. You will be taken off study if intolerable side effects occur or if you are unable to follow study directions.

Follow-Up:

Thirty (30) days after your study visit you will be called by the study staff and asked how you are feeling and about any side effects you may be having. This call should last about 10 minutes.

This is an investigational study. Fentanyl is FDA approved and commercially available for the treatment of pain. Its use to control shortness of breath is investigational.

Up to 20 participants will be enrolled in this study. All will take part at MD Anderson.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of cancer with evidence of active disease
2. Breakthrough dyspnea, defined in this study as dyspnea on exertion with an average intensity level >/=3/10 on the numeric rating scale
3. Outpatient at MD Anderson Cancer Center seen by the Supportive Care Service, Thoracic Medical Oncology or Cardiopulmonary Center
4. Ambulatory and able to walk with or without walking aid
5. On strong opioids with morphine equivalent daily dose of 60-130 mg for at least one week, with stable (i.e. +/- 30%) regular dose over the last 24 hours
6. Karnofsky performance status >/=50%
7. Age 18 or older
8. Able to complete study assessments
9. Must speak and understand English.

Exclusion Criteria:

1. Dyspnea at rest >/=7/10 at the time of enrollment
2. Supplemental oxygen requirement >6 L per minute
3. Delirium (i.e. Memorial delirium rating scale >13)
4. History of unstable angina or myocardial infarction 1 month prior to study enrollment
5. Resting heart rate >120 at the time of study enrollment
6. Systolic pressure >180 mmHg or diastolic pressure >100 mmHg at the time of study enrollment
7. History of active opioid abuse within the past 12 months
8. History of allergy to fentanyl
9. Severe anemia (Hb <7g/L) if documented in the last month and not corrected prior to study enrollment*
10. Bilirubin >5X Upper limit of normal if documented in the last month and not lowered to <5x normal prior to study enrollment*
11. Diagnosis of acute pulmonary embolism within past 2 weeks
12. Diagnosis of pulmonary hypertension
13. Unwilling to provide informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2014-05-27 (Actual); Primary Completion 2019-12-04 (Actual); Study Completion 2019-12-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David Hui, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- University of Texas MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: University of Texas MD Anderson Cancer Center Website — http://www.mdanderson.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Adult participants (age>18) with an active diagnosis of cancer were recruited between May 2014 to May 2016 from the Supportive Care Center outpatient clinic of MD Anderson Cancer Center who met the inclusion and exclusion criteria.
Pre-assignment Details: A total of 36 participants enrolled. 22 patients were randomized, 14 patients dropped out before randomization, 3 participants died, 4 had declining Karnofsky Performance Score/hospice, 2 participant's Morphine equivalent daily dose was no longer in range, 1 participant declined and 4 participants were no longer interested in the study.
Groups:
- Intervention Group (Fentanyl Buccal Tablet): Received Fentanyl Buccal Tablet 30 minutes before 2nd 6 minute walk test, dose equivalent to 20-50% of their total opioid dose over the past 24 hours.
- Controlled Group (Placebo): Received Placebo tablet 30 minutes before 2nd 6 minute walk test.
Period: Overall Study
Arm/Group | Intervention Group (Fentanyl Buccal Tablet) | Controlled Group (Placebo)
Started | 11 | 11
Completed | 9 | 11
Not Completed | 2 | 0
Not completed — Withdrawal by Subject | 1 | 0
Not completed — Adverse Event | 1 | 0

BASELINE CHARACTERISTICS:
Population: The data provided is for the 20 participants that completed the study.
Groups:
- Total: Total of all reporting groups
Arm/Group | Intervention Group (Fentanyl Buccal Tablet) | Controlled Group (Placebo) | Total
Number analyzed (Participants) | 9 | 11 | 20
Age, Continuous [Mean (Full Range); unit: years] | 52 [31 to 67] | 57 [45 to 72] | 55 [31 to 72]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 6 | 12
  Male | 3 | 5 | 8
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 2 | 2
  Not Hispanic or Latino | 9 | 9 | 18
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 3 | 5
  White | 7 | 8 | 15
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 9 | 11 | 20
Education [Count of Participants; unit: Participants]
  High School or less | 7 | 9 | 16
  College and above | 2 | 2 | 4
Cancer Stage [Count of Participants; unit: Participants]
  Metastatic Stage | 9 | 10 | 19
  Locally Advanced | 0 | 1 | 1
Cancer Type [Count of Participants; unit: Participants]
  Lung Cancer | 3 | 5 | 8
  Breast Cancer | 1 | 2 | 3
  Gastrointestinal Cancer | 2 | 1 | 3
  Genitourinary Cancer | 2 | 1 | 3
  Other | 1 | 1 | 2
  Gynecologic Cancer | 0 | 1 | 1

OUTCOME MEASURES:

1. Primary Outcome: Dyspnea Numeric Rating Scale
Description: Our primary outcome was dyspnea intensity "now" using a dyspnea numeric rating scale that ranges from 0 ("no shortness of breath") to 10 ("worst possible shortness of breath"). Measured the mean difference between the baseline and second 6 minute walk test. 6 minute walk tests were carried out following guidelines from the American Thoracic Society.
Time Frame: Baseline to 30 minutes
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Intervention Group (Fentanyl Buccal Tablet) | Controlled Group (Placebo)
Number analyzed (Participants) | 9 | 11
score on a scale | -2.4 [-3.5 to -1.3] | -1.1 [-2.5 to 0.2]

2. Secondary Outcome: Dyspnea Borg Scale
Description: Assessed dyspnea using the 0-10 modified Dyspnea Borg Scale at baseline walk test and after second 6 minute walk test. The Borg scale ranges from 0 ("no shortness of breath") to 10 ("worst possible shortness of breath"). Measured the mean difference between the baseline walk test and second 6 minute walk test.
Time Frame: Baseline to 30 minutes
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Intervention Group (Fentanyl Buccal Tablet) | Controlled Group (Placebo)
Number analyzed (Participants) | 9 | 11
score on a scale | -1.6 [-2.9 to -0.3] | -0.5 [-1.9 to 0.8]

3. Secondary Outcome: Walk Distance at 6 Minutes
Description: Measured the mean difference between the baseline walk test and second 6 minute walk test.
Time Frame: Baseline to 30 minutes
Measure: Mean (95% Confidence Interval); unit: meters
Arm/Group | Intervention Group (Fentanyl Buccal Tablet) | Controlled Group (Placebo)
Number analyzed (Participants) | 9 | 11
meters | -1 [-22.3 to 20.3] | 6.7 [-3.4 to 16.9]

ADVERSE EVENTS:
Time Frame: Each adverse effect was measured using an 11-point numeric rating scale (0=none, 10=worst) immediate before drug administration and immediately after the second 6 minute walk test (approximately 30 minutes later).
Groups:
- Controlled Group (Placebo): Received Placebo tablet 30 minutes before 2nd 6 minute walk test.
  .
Arm/Group | Intervention Group (Fentanyl Buccal Tablet) | Controlled Group (Placebo)
All-Cause Mortality (participants affected / at risk) | 0/9 | 0/11
Serious Adverse Events (participants affected / at risk) | 0/9 | 0/11
Other Adverse Events (participants affected / at risk) | 0/9 | 2/11
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Intervention Group (Fentanyl Buccal Tablet) (N=9) | Controlled Group (Placebo) (N=11)
Dizzy (Nervous system disorders) | 0 | 2
Drowsy (Nervous system disorders) | 0 | 2
Itchiness (Skin and subcutaneous tissue disorders) | 0 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-03-08): https://cdn.clinicaltrials.gov/large-docs/14/NCT01856114/Prot_SAP_000.pdf